CLINICAL TRIAL: NCT02808624
Title: The Potential Prophylactic Effect of Exogenous Antioxidant ''L-CARNOSINE'' on Oxaliplatin-induced Peripheral Neuropathy in Cancer Patients
Brief Title: L-carnosine Prophylactic Effect on Oxaliplatin Induced Peripheral Neuropathy in GIT Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Misr International University (Other); Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Magdy, Teaching assistant, Misr International University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PT(1451)
Record Dates: First submitted 2016-05-20; First posted 2016-06-22 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Neuropathy; Cancer
Keywords: Oxaliplatin, peripheral neuropathy, L-CARNOSINE
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neoplasms | interventions — Carnosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): this arm will receive L-CARNOSINE PO (each patient will receive 1 tablet daily and each tablet contains 500 mg thus a total of 500 mg per day) together with their chemotherapy wich is oxaliplatin.
  Interventions: Drug: L-CARNOSINE
- Control group (No Intervention): This arm wont receive L-CARNOSINE, they will receive their chemotherapy (oxaliplatin) only.

INTERVENTIONS:
Drug: L-CARNOSINE — L-CARNOSINE is a supplement given with chemotherapy to prevent peripheral neuropathy.
  Other Names: CARNOSINE
  Arms: Treatment group

SUMMARY:
This study evaluates the prophylactic effect of exogenous L-CARNOSINE in Oxaliplatin induced peripheral neuropathy, Thus half of the patients will receive L-CARNOSINE with Oxaliplatin and the other half will not receive L-CARNOSINE with their chemotherapy (oxaliplatin),And then neuropathy together with some oxidative stress markers will be assessed at the end of treatment duration (three months) .

DETAILED DESCRIPTION:
Oxaliplatin causes peripheral neuropathy , L-CARNOSINE is supposed to prevent this side effect possibly by reducing oxidative stress and enhancing the growth of nerves.This study is intended to clarify the effect and mechanism of action of L-CARNOSINE in preventing Oxaliplatin induced peripheral neuropathy in cancer patients.

Blood samples will be collected from the patients before starting the chemotherapy and at the end of treatment duration (3 months) and then oxidative stress markers will be measured in these samples

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be enrolled in this study, if they meet the following criteria

1. Elderly males and females with age (˃18 and ˂60).
2. Cancer patients treated with oxaliplatin for the first time (dose 85- 135mg/m2) administered every two to three weeks for 3 months.

Exclusion Criteria:

Excluded from this study are the patients with the following Criteria:

* Suffering from diabetes mellitus.
* Suffering from peripheral neuropathy as a result of any other disease or drug.
* Suffering from severe renal impairment (CrCl ˂ 30 ml/min).
* Suffering from epilepsy.
* Taking vitamin B.
* Who previously took Oxaliplatin or any other chemotherapeutic agent that causes peripheral neuropathy.
* Taking antidepressants or MAOI's.
* Taking NSAIDs, paracetamol, opiates or any other analgesics or pain killers.
* Pregnant or lactating patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessment of peripheral neuropathy using neuropathy grading score "CTCAE", version 4.0) also oxidative stress markers will be measured by ELISA kits. | Three months
  The following markers will be measured by ELISA kits :
  Nrf2 induced oxidative stress pathways (GSH) NF-KB anti-inflammatory pathway (TNF- alpha) pro-apoptic signals (caspase 3)

SECONDARY OUTCOMES:
Assessment of tumor markers (CA,CEA) in blood. | Three months
  Tumor Markers (CA,CEA) will be assessed at the end of treatment duration to make sure that L-CARNOSINE didn't interfere with the patients' response to chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Samira Saleh, Professor, Study Director — Cairo University; Hanan elabhar, Professor, Study Chair — Cairo University; Mona Schaalan, assoc. prof., Study Chair — Misr International University; Amr Shafik, Assoc. Prof, Study Chair — Ain Shams University
Locations (1):
- Cairo University, Cairo, Kasr El Aini, Egypt